CLINICAL TRIAL: NCT02943161
Title: Asthma L-Citrulline Pilot Study
Acronym: ALPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2041
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Asthma
Keywords: Obesity; L-citrulline
MeSH Terms: conditions — Asthma; Obesity | interventions — Citrulline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-Citrulline (Experimental): In this pilot study subjects with asthma that have an increased body mass index compatible with being obese, will be invited to participate in a short open-label treatment with 15g/day of L-citrulline for two weeks. Study participants will be asked to do lung function testing and donate blood before and after taking the supplement. L-citrulline is safe and well tolerated and has been used at much higher doses without significant side effects.
  Interventions: Dietary Supplement: L-Citrulline

INTERVENTIONS:
Dietary Supplement: L-Citrulline — The purpose of this study is to see if citrulline supplementation will restore NO levels and lung function in subjects with asthma.

SUMMARY:
This study will evaluate whether treatment with L-citrulline, which is an amino acid found in some foods, can increase levels of L-arginine and thereby restore the concentration of nitric oxide (NO) in the airways.

DETAILED DESCRIPTION:
Research has shown that some obese asthmatics have a metabolic imbalance in which L-arginine levels are reduced. L-arginine is an amino acid that is used to make NO, a gas that is normally made in the bronchi and ensures that the lungs function properly. In this pilot study subjects with asthma that have an increased body mass index compatible with being obese, will be invited to participate in a short open-label treatment with 15g/day of L-citrulline for two weeks. Study participants will be asked to do lung function testing and donate blood before and after taking the supplement. L-citrulline is safe and well tolerated and has been used at much higher doses without significant side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adequate completion of informed consent process with written documentation
* Male and female patients, 18 - 70 years old, inclusive
* Physician diagnosis of asthma (for medical records, ICD 10 coding for physician's diagnosis)
* All racial/ethnic backgrounds may participate
* BMI ≥ 30
* Treatment of controller asthma medication(s) ≥ 4 weeks
* Smoking history ≤10 pack years and no smoking in the last year
* V1 eNO ≤ 30ppb (may be repeated 3x during visit; lowest ppb will be kept)

Exclusion Criteria:

* Respiratory tract infection within the 4 weeks prior to the study (may re-enroll after 4 weeks).
* Oral or systemic corticosteroid burst (for any indication) within the 4 weeks
* One-time doses, such as intra-articular injections into a shoulder or knee joint, require a 2-week washout.
* Asthma-related ER visit within the previous 4 weeks of Visit 1
* Significant concomitant medical illness, including (but not limited to)

  * Heart disease
  * Cancer
  * Uncontrolled diabetes,
* Chronic renal failure (creatinine > 2.0) at Visit 1 (Associated with higher ADMA levels)
* Untreated sleep apnea
* Other chronic lung/respiratory diseases (COPD, IPF, etc.)
* High dose inhaled steroids (> 1000 mcg/day of Fluticasone or equivalent)
* Current statin use (statins lower ADMA levels); patients may stop statins with approval from their primary physician and enroll after a 6-week washout
* Positive urine pregnancy test at Visit 1 or at any time during the study
* Intolerance or allergy to L-arginine or L-citrulline
* Concomitant use of PDE5 drugs or oral mononitrates
* Participation in an intervention study, use of investigative drugs within the past 30 days or plans to enroll in such a trial during the study
* Unable or unlikely to complete study assessments in the opinion of the Investigator
* Study intervention poses undue risk to patient in the opinion of the Investigator
* Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Exhaled Nitric Oxide (eNO) | 2 weeks or 14 days
  Change in eNO levels before and after treatment with open label L-citrulline at 15g/day

SECONDARY OUTCOMES:
Change in Plasma L-arginine/ADMA Ratio | 2 weeks or 14 days
  Change in L-arginine/ADMA before and after 2 weeks of L-citrulline at 15g/day

OTHER OUTCOMES:
Change in Asthma Control Score | 2 weeks or 14 days
  Change in asthma control scores (ACQ)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Sharing de-identified data with co-investigators approved by the IRB and Duke University